CLINICAL TRIAL: NCT00255411
Title: Neuropsychiatric Correlates of Psychogenic Movement Disorder and Non-Epileptic Seizure
Brief Title: Psychiatric Correlates of Psychogenic Movement Disorder and Non-Epileptic Seizure
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060027; 06-N-0027
Record Dates: First submitted 2005-11-17; First posted 2005-11-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-02-24

CONDITIONS: Psychogenic Movement Disorders; Non-epileptic Seizures
Keywords: Conversion Disorder; Somatoform Disorder; Involuntary Movement; Childhood Abuse; Depression; Psychogenic Movement Disorder; PMD; Non-Epileptic Seizure; NES; Healthy Volunteer; HV
MeSH Terms: conditions — Seizures; Conversion Disorder; Somatoform Disorders; Dyskinesias; Depression

SUMMARY:
This study will explore how the mind and the brain work to cause movement symptoms or seizures in people who do not have a recognized neurological or medical disorder. The study includes a check for psychiatric disorders, symptoms and their severity; psychiatric and personality questionnaires; and neuropsychological testing.

Normal, healthy volunteers, people who have movement symptoms not due to a brain or medical disorder and people who have seizures not due to epilepsy may be eligible for this study. All candidates must be 18 years of age or older.

All participants have a medical history, physical examination and psychological evaluation, including completion of questionnaires. People with movement symptoms or seizures have a symptoms evaluation.

Some participants also undergo neuropsychological testing, including questionnaires, pen-and-paper or computerized tests, and motor tasks.

DETAILED DESCRIPTION:
Objectives

The objectives of this study are (1) to investigate the relationship between childhood abuse and dissociative experiences in both psychogenic movement disorders (PMD) and non-epileptic seizures (NES) and (2) to investigate the relationship between childhood abuse and both PMD and NES. The secondary objective of the study is to investigate if measures of response inhibition differ between PMD subjects compared to normal controls. This study is part of a larger study investigating the psychological and biological correlates of conversion disorder.

Study population

We intend to study adult patients with diagnoses of PMD seen by the Human Motor Control Section clinic or patients with diagnoses of NES seen by the Epilepsy clinic and normal controls.

Design

A psychiatric assessment, measurement scales and neuropsychological testing will be administered to the PMD and NES patients and normal controls.

Outcome measures

The first primary outcome measure will be the comparison of the different subtypes of childhood abuse (as measured by the Childhood Trauma Interview) and the severity of dissociation (as measured by the Dissociative Experiences Scale). The second primary outcome measure will be the comparison of frequencies of different subtypes of childhood abuse (as measured by the Childhood Trauma Interview) between PMD, NES and normal control groups. The secondary outcome measure will be the comparison of stop-signal reaction time as measured with the stop-signal task.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients for dissociation study:

* Diagnosis of clinically definite PMD utilizing Fahn and Williams criteria. The diagnosis will be made by a movement disorders neurologist.
* Or a diagnosis of NES based on video-EEG. The diagnosis will be made by an epileptologist.
* Males or females
* Age 18 or older
* Able to provide informed consent

Patients for cognitive study:

* Diagnosis of clinically definite PMD utilizing Fahn and Williams criteria. The diagnosis will be made by a movement disorders neurologist.
* Age 18 or older
* Males or females
* Able to provide informed consent

Normal volunteers for cognitive study:

* Normal volunteers age 18 or older will be included
* Males or females
* Able to provide informed consent

EXCLUSION CRITERIA:

Patients for dissociation study:

* Diagnosis of probable or possible PMD using Fahn and Williams criteria.
* Patients with neurological disorders with elaboration of their underlying disease process including comorbid epilepsy.
* Patients with a medical condition that prevents them from taking part in the study.
* Patients with current suicidal ideation.
* Patients with a psychotic disorder.
* Patients with active substance abuse within the last 6 months.
* Patients below the age of 18.
* Patients who are not capable of consent.
* Patients with an IQ less than 55.
* Patients currently involved in lawsuits.

Patients for cognitive study:

* Diagnosis of probable or possible PMD using Fahn and Williams criteria
* Patients with neurological disorders with elaboration of their underlying disease process including comorbid epilepsy
* Patients with a medical condition that prevents them from taking part in the study.
* Patients with a history of a neurological disorder (e.g. dementia, cerebrovascular accident, neurodegenerative disorder, inflammatory disorders or infections of the central nervous system) that may result in cognitive deficits.
* Patients with a history of traumatic brain injury resulting in loss of consciousness or amnesia lasting for more than a few seconds.
* Patients with a psychotic disorder or bipolar disorder
* Patients with a current major depression
* Patients with current moderate to severe anxiety (Hamilton Anxiety Rating Scale greater than 25)
* Patients with current attention deficit hyperactivity disorder.
* Patients with active substance abuse within the last 6 months.
* Patient with current suicidal ideation.
* Patients below the age of 18.
* Patients who are not capable of consent.
* Patients with an IQ less than 55.
* Patients currently involved in lawsuits.

Normal volunteers for cognitive study:

* Normal volunteers younger than 18 years
* Normal volunteers with an active medical condition that might prevent participation.
* Normal volunteers with a history of neurological disorders (e.g. dementia, cerebrovascular accident, neurodegenerative disorder, inflammatory disorders or infections of the central nervous system) that may result in cognitive deficits
* Normal volunteers with a history of traumatic brain injury resulting in loss of consciousness or amnesia lasting for more than a few seconds
* Normal volunteers with a psychotic disorder or bipolar disorder
* Normal volunteers with a current major depression
* Normal volunteers with moderate to severe anxiety (Hamilton Anxiety Rating Scale greater than 25)
* Normal volunteers with active substance abuse within the last 6 months
* Normal volunteers with current attention deficit hyperactivity disorder
* Normal volunteers with an IQ less than 55
* Normal volunteers who are not capable of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190
Dates: Start 2005-11-09; Study Completion 2009-02-24

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Williams DT, Ford B, Fahn S. Phenomenology and psychopathology related to psychogenic movement disorders. Adv Neurol. 1995;65:231-57. No abstract available. PMID 7872143
- [Background] Carson AJ, Ringbauer B, Stone J, McKenzie L, Warlow C, Sharpe M. Do medically unexplained symptoms matter? A prospective cohort study of 300 new referrals to neurology outpatient clinics. J Neurol Neurosurg Psychiatry. 2000 Feb;68(2):207-10. doi: 10.1136/jnnp.68.2.207. PMID 10644789
- [Background] Stone J, Carson A, Sharpe M. Functional symptoms and signs in neurology: assessment and diagnosis. J Neurol Neurosurg Psychiatry. 2005 Mar;76 Suppl 1(Suppl 1):i2-12. doi: 10.1136/jnnp.2004.061655. No abstract available. PMID 15718217